CLINICAL TRIAL: NCT03967964
Title: Prospective, Randomized, Open-label and Comparative Study to Determine the Pharmacokinetic Parameters of Vaginal Rings That Contain DHEA, Testosterone, or the Combination of Both Androgens, in Comparison With Oral Administration of DHEA and Transdermal Administration of Testosterone, in Postmenopausal Women
Brief Title: Pharmacokinetics of a Novel Vaginal Delivery System for Testosterone and Dehydroepiandrosterone (DHEA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Andromaco S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKAVD+T; EC1503 (Other: Sponsor code)
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Pharmacokinetics; Hormone Deficiency
Keywords: Gynaecology; Obstetrics
MeSH Terms: interventions — Dehydroepiandrosterone; Testosterone

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, open-label comparative, single-site study with 5 treatment groups. Each participant receives a single Treatment for 72 hours. Allocation to Treatment is in a 1:1:1:1:1 order.

ARMS (5):
- Group 1: AVD (Experimental): Vaginal ring with 2.2 grams dehydroepiandrosterone (DHEA), wearing time 72 hours
  Interventions: Drug: Dehydroepiandrosterone 2.2 g
- Group 2: AVT (Experimental): Vaginal ring with 35 mg testosterone, wearing time 72 hours.
  Interventions: Drug: Testosterone
- Group 3: AVD+T (Experimental): Vaginal ring with 1.5 grams DHEA and 25 mg testosterone, wearing time 72 hours.
  Interventions: Drug: Dehydroepiandrosterone 1.5 g/Testosterone 25 mg
- Group 4: DHEA capsule (Active Comparator): Capsules with 25 mg DHEA, oral administration every 8 hours for a 72-hour period.
  Interventions: Drug: Dehydroepiandrosterone Oral Capsule
- Group 5: Testosterone transdermal gel (Active Comparator): Testosterone transdermal gel with dosing valve (pump): administration of 3 pump actuations (equivalent to 5 mg of testosterone each) per day (total daily dose 15 mg), on 3 consecutive days (72 hours).
  Interventions: Drug: Testosterone Topical Gel

INTERVENTIONS:
Drug: Dehydroepiandrosterone 2.2 g — Vaginal ring with 2.2 grams DHEA.
  Arms: Group 1: AVD
Drug: Dehydroepiandrosterone 1.5 g/Testosterone 25 mg — Vaginal ring with DHEA 1.5 grams/Testosterone 25 mg.
  Arms: Group 3: AVD+T
Drug: Testosterone — Vaginal ring with 35 mg testosterone.
  Arms: Group 2: AVT
Drug: Testosterone Topical Gel — Gel containing 1% testosterone.
  Other Names: ActiserPump®
  Arms: Group 5: Testosterone transdermal gel
Drug: Dehydroepiandrosterone Oral Capsule — Capsule containing 25 mg DHEA
  Arms: Group 4: DHEA capsule

SUMMARY:
This study was performed to determine the pharmacokinetic parameters of vaginal rings that contain DHEA, testosterone, or combinations of both androgens, in comparison to the oral administration of DHEA and the transdermal administration of testosterone.

ELIGIBILITY:
Inclusion Criteria:

* Women between 40 to 60 years old.
* Postmenopausal with spontaneous amenorrhea of 1 year or more, regardless of follicle stimulating hormone (FSH) levels; or amenorrhea of 6 to 12 months, in which the postmenopausal state will be confirmed with a FSH level of 0.040 international units per milliliter or higher.
* Body Mass Index between 19 and 30.
* Intact uterus.
* Not having received hormone therapy in the month prior to selection.
* Adequate veins to conduct serial blood samplings.
* Recent Pap smear (not more than 12 months), with a result negative for malignant neoplastic cells, and that contains sufficient endocervical cells for analysis. If the Pap smear was performed more than 12 months ago or cannot be verified through clinical documentation, it must be repeated during the selection process.
* Normal mammogram, BI.RADS I or II (American College of Radiology), within the last year. If the mammogram was performed more than 12 months ago or cannot be verified through clinical documentation, it must be repeated during the selection process.
* That provide written informed consent.

Exclusion Criteria:

* Use at randomization of phenytoin, barbiturates, primidone, carbamazepine, rifampin, griseofulvin, ketoconazole, lipid-lowering agents.
* History of diseases such as coronary heart disease, breast cancer, uterine cancer, and/or chronic hepatic disease.
* Unconscious volunteers, severely ill, or with mental disability.
* Allergy and hypersensitivity to DHEA and/or testosterone.
* Untreated or uncontrolled hypertension, with systolic pressure above 140 mm Hg or diastolic pressure above 90 mm Hg.
* Current participation in other research at the moment of the screening visit, or having concluded their participation in a previous research in less than 30 days since their last visit.
* Pregnant or lactating women; pregnancy must be confirmed with a urine positive human chorionic gonadotropin (HCG) test during screening.
* History of vein thrombosis (deep vein thrombosis, pulmonary embolism).
* History of arterial thrombosis (myocardial infarction) or prodromic conditions (e.g. transient ischemic attack, angina pectoris).
* History of stroke.
* History of migraine with focal neurological manifestations.
* History of hepatic tumor (benign or malignant).
* History of clinical atherosclerosis in first grade relatives (parents, siblings, sons [men less than 55 years old and women less than 65 years old]).
* Smoking (5 or more cigarettes a day).
* Diabetes mellitus that will be ruled out at screening if fasting glucose is less than 100 mg/dL or between 100 and 125 mg/dL, with Oral Glucose Tolerance Test that rules out diabetes. Diabetes will be confirmed with blood glucose equal to or above 200 mg/dL or 2 fasting glucose tests equal to or above 126 mg/dL.
* High density lipopolysaccharide (HDL)-cholesterol below 35 mg/dL.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2016-07-15 (Actual); Study Completion 2016-07-15 (Actual)

PRIMARY OUTCOMES:
Testosterone: Area under the serum concentration time curve (AUC0-72) | Pre-dose and from 30 minutes after administration of the assigned treatment to 72 hours
  Serum testosterone was measured pre-dose and at 30 minutes, at 1 hour, 2, 4, 6, 8, 24, 48, and 72 hours after vaginal ring insertion, the transdermal application of the testosterone gel, or after taking DHEA capsules. The AUC0-72 was calculated.
DHEA: Area under the serum concentration time curve (AUC0-72) | Pre-dose and from 30 minutes after administration of the assigned treatment to 72 hours
  Serum DHEA were measured pre-dose and at 30 minutes, at 1 hour, 2, 4, 6, 8, 24, 48, and 72 hours after vaginal ring insertion, the transdermal application of the testosterone gel, or after taking DHEA capsules. The AUC0-72 was calculated.
Testosterone: Average serum concentration 0-24 hours | Pre-dose and from 30 minutes after administration of the assigned treatment to 24 hours
  Serum testosterone was measured pre-dose and at 30 minutes, at 1 hour, 2, 4, 6, 8, 24, 48, and 72 hours after vaginal ring insertion, the transdermal application of the testosterone gel, or after taking DHEA capsules. The average serum concentration achieved in the first 24 hours after administration of the assigned treatment was calculated.
DHEA: Average serum concentration 0-24 hours | Pre-dose and from 30 minutes after administration of the assigned treatment to 24 hours
  Serum DHEA was measured pre-dose and at 30 minutes, at 1 hour, 2, 4, 6, 8, 24, 48, and 72 hours after vaginal ring insertion, the transdermal application of the testosterone gel, or after taking DHEA capsules. The average serum concentration achieved in the first 24 hours after administration of the assigned treatment was calculated.
Testosterone: Maximum serum concentration (Cmax) | Pre-dose and from 30 minutes after administration of the assigned treatment to 72 hours
  Serum testosterone was measured pre-dose and at 30 minutes, at 1 hour, 2, 4, 6, 8, 24, 48, and 72 hours after vaginal ring insertion, the transdermal application of the testosterone gel, or after taking DHEA capsules. Cmax was calculated.
DHEA: Maximum serum concentration (Cmax) | Pre-dose and from 30 minutes after administration of the assigned treatment to 72 hours
  Serum DHEA was measured pre-dose and at 30 minutes, at 1 hour, 2, 4, 6, 8, 24, 48, and 72 hours after vaginal ring insertion, the transdermal application of the testosterone gel, or after taking DHEA capsules. Cmax was calculated.
Testosterone: Time to achieve maximum serum concentration (tmax) | pre-dose and from 30 minutes after administration of the assigned treatment to 72 hours
  Serum testosterone was measured pre-dose and at 30 minutes, at 1 hour, 2, 4, 6, 8, 24, 48, and 72 hours after vaginal ring insertion, the transdermal application of the testosterone gel, or after taking DHEA capsules. Tmax was calculated.
DHEA: Time to achieve maximum serum concentration (tmax) | pre-dose and from 30 minutes after administration of the assigned treatment to 72 hours
  Serum DHEA was measured pre-dose and at 30 minutes, at 1 hour, 2, 4, 6, 8, 24, 48, and 72 hours after vaginal ring insertion, the transdermal application of the testosterone gel, or after taking DHEA capsules. Tmax was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (1):
- Instituto de Investigación Materno Infantil (IDIMI) - Maternidad Hospital San Borja (HCSBA), Santiago, Chile

IPD SHARING:
Plan to Share IPD: No